CLINICAL TRIAL: NCT05851066
Title: A Phase 1 Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of VSA003 in Chinese Adult Healthy Volunteers
Brief Title: A VSA003 Phase 1 Study in Chinese Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Visirna Therapeutics HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VSA003-1001
Record Dates: First submitted 2023-04-26; First posted 2023-05-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Dyslipidemias; Familial Hypercholesterolemia; Hypertriglyceridemia
MeSH Terms: conditions — Dyslipidemias; Hyperlipoproteinemia Type II; Hypertriglyceridemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VSA003 (Experimental): single dose of VSA003 by subcutaneous (sc) injections: 50 mg, 100 mg, 200 mg
  Interventions: Drug: VSA003
- placebo (Placebo Comparator): sterile normal saline (0.9% NaCl) calculated volume to match active treatment
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: VSA003 — sequential dosing, SC, single dose: 50 mg, 100 mg, 200 mg
  Arms: VSA003
Drug: 0.9% NaCl — placebo
  Arms: placebo

SUMMARY:
This is a randomized, double blinded, phase 1 study. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single dose of VSA003 in healthy adult volunteerst

ELIGIBILITY:
Inclusion Criteria:

* Women of child bearing potential must have a negative pregnancy test, cannot be breastfeeding and must be willing to use contraception
* BMI 18.0~28.0 kg/m2
* Willing to provide written informed consent and to comply with study requirements
* On a stable diet for at least 4 weeks with no plans to significantly alter diet or weight over course of study
* TG> 100 mg/dL
* LDL-C> 70 mg/dL

Exclusion Criteria:

* Clinically significant health concerns
* Regular use of alcohol within one month prior to screening
* Recent (within 3 months) use of illicit drugs
* Female with pregnancy or breastfeeding
* QTcF>450 ms in ECG
* Donation or loss of whole blood more than 400 ml prior to administration of the study treatment

Note: additional inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse event (AE) and serious adverse event (SAE) | Up to 85±3 days post-dose
  safety and tolerability

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of VSA003 | Up to 48 hours post dose
  pharmacokinetics (PK)
Time of occurrence of Cmax (tmax) of VSA003 | Up to 48 hours post dose
  PK
Apparent terminal phase half-life (t1/2) of VSA003 | Up to 48 hours post dose
  PK
Area under the concentration-time curve from time zero (pre-dose) to the last quantifiable concentration (AUC0-t) of VSA003 | Up to 48 hours post dose
  PK
Apparent clearance (CL/F) of VSA003 | Up to 48 hours post dose
  PK
Apparent terminal phase volume of distribution (Vz/F) of VSA003 | Up to 48 hours post dose
  PK
Change of fasting serum ANGPTL3 from pre-dose baseline | Up to 85±3 days post-dose
  PD
Anti-drug Antibodies (ADA) to VSA003 | Up to 85±3 days post-dose
  immunogenecity

OTHER OUTCOMES:
Change of low density lipoprotein cholesterol (LDL-C) from pre-dose baseline | Up to 85±3 days post-dose
  Lipid profile
Change of total cholesterol (TC) from pre-dose baseline | Up to 85±3 days post-dose
  Lipid profile
Change of triglyceride (TG) from pre-dose baseline | Up to 85±3 days post-dose
  Lipid profile
Change of high density lipoprotein cholesterol (HDL-C) from pre-dose baseline | Up to 85±3 days post-dose
  Lipid profile
Change of fasting glucose from pre-dose baseline | Up to 85±3 days post-dose
  glucose metabolism
Change of HbA1c from pre-dose baseline | Up to 85±3 days post-dose
  glucose metabolism
Change of fasting C peptide from pre-dose baseline | Up to 85±3 days post-dose
  glucose metabolism
Change of fasting insulin from pre-dose baseline | Up to 85±3 days post-dose
  glucose metabolism

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No